CLINICAL TRIAL: NCT02831400
Title: Changes in Circulatory I-FABP in Elderly Persons in Daily Life: A Pilot Study
Brief Title: Changes in Circulatory I-FABP in Elderly Persons in Daily Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Suzanne Stokmans, MD, PhD candidate, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL54574.042.16
Record Dates: First submitted 2016-07-07; First posted 2016-07-13 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Malnutrition; Intestinal Integrity; Intestinal Fatty Acid Binding Protein (IFABP)
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFABP assessment (1 study group) (Experimental): 30 elderly volunteers
  Interventions: Behavioral: Walking test; Behavioral: Standard Meal

INTERVENTIONS:
Behavioral: Walking test — Walking test to increase cardiac output, maximum 12 minutes
Behavioral: Standard Meal — After the walking test, volunteers eat a standard warm meal

SUMMARY:
The purpose of this study is to detect changes in circulatory I-FABP values (50% increase) in elderly volunteers following the combination of moderate physical activity and a standard meal.

ELIGIBILITY:
Inclusion Criteria:

1. Age 75 years or older (both sexes)
2. Participating in the Embrace project.

Exclusion Criteria:

1. Previous gastrointestinal resections
2. Chronic inflammatory gastrointestinal disease

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
50% increase of I-FABP in plasma. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: BL van Leeuwen, MD, PhD, Principal Investigator — University Medical Center Groningen; JJ de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No